CLINICAL TRIAL: NCT05379270
Title: Intergenerational Transmission of Low-calorie Sweeteners Via Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NCR213471
Record Dates: First submitted 2022-05-11; First posted 2022-05-18 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Breastfeeding
Keywords: low-calorie sweeteners; sucralose; acesulfame-potassium; pharmacokinetics; breast milk; lactation
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diet soda (Experimental): Participants will be asked to ingest 24 of a commercially-available diet beverage sweetened with sucralose and acesulfame-potassium.
  Interventions: Other: Diet soda

INTERVENTIONS:
Other: Diet soda — Participants will be asked to drink 24 ounces of a commercially-available diet beverage sweetened with sucralose and acesulfame-potassium.

SUMMARY:
This project aims to measure the widely consumed low-calorie sweeteners (LCS) sucralose and acesulfame-potassium, in maternal breast milk and plasma at pre-specified timepoints over 72 hours and in a single sample of infants' plasma. Sucralose and acesulfame-potassium concentrations will be measured using liquid chromatography-mass spectrometry (LC-MS). The data generated will inform the design of larger, longer-term, prospective studies needed to investigate clinically-relevant consequences of early life LCS exposure in humans.

DETAILED DESCRIPTION:
Low-calorie sweetener (LCS) consumption is highly prevalent among lactating women, yet the current understanding of LCS effects on diet, weight, and health is extremely limited, especially when exposure begins early in life. This project aims to measure the widely consumed LCSs, sucralose and acesulfame-potassium, in maternal breast milk and plasma, at pre-specified, time-points over the course of 72 hours, and in a single sample of infants' plasma (analyzed using a population pharmacokinetics approach).

Mothers will attend an enrollment visit, which will take place virtually and will schedule an in-person visit to take place at Children's National Hospital approximately one week later. During the enrollment visit, informed consent will be obtained and demographic, anthropometric, and dietary data will be collected. During the week prior to their scheduled in-person study visit, mothers will be instructed to continue their usual dietary habits and to complete an online, photo-assisted, 7-day food record.

Mothers will be instructed to arrive fasted for the in-person visit, which will last for approximately 13 hours. Following ingestion of a diet beverage containing sucralose and ace-K, mothers will remain at Children's National for supervised serial sample collection at pre-determined time points over 12 hours, and will provide additional samples on three subsequent consecutive days (72 hours). Mothers will be instructed to continue to complete the online, photo-assisted, food record for the three days following the in-person study visit (until 72 hours following diet beverage consumption).

A plasma sample will be collected from each infant via heel-stick at one of the following pre-specified time intervals following the mother's ingestion of the diet beverage: 1.5-3 hours, 3-5 hours, 5-7 hours, 7-9 hours, 9-14 hours, and 22-36 hours.

ELIGIBILITY:
Inclusion Criteria:

* mother gave birth within the past 6 months
* mother ≥18 years of age
* exclusively breastfeeding
* reports consumption of diet, low-calorie sweetener-containing beverages ≥ 1 time per week.
* infants' corrected age >= 4 weeks

Exclusion Criteria:

* known allergy or contraindication to sucralose or acesulfame-potassium (infant or mother)
* active nutritional disorder known to cause malabsorption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2022-12-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Sylvetsky AC, Kuttamperoor JT, Langevin B, Murphy J, Arcaro KF, Smolyak S, Walter PJ, Cai H, Daines DH, van den Anker JN, Gopalakrishnan M. Intergenerational transmission of sucralose and acesulfame-potassium from mothers to their infants via human milk: a pharmacokinetic study. Am J Clin Nutr. 2024 Oct;120(4):846-853. doi: 10.1016/j.ajcnut.2024.08.001. Epub 2024 Aug 5. PMID 39111550

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mother-infant dyads are recruited between February 2022 and November 2022 at the George Washington University Medical Faculty Associates Obstetrics & Gynecology clinic, using the clinic-based mobile application Babyscripts, as well as through local social media and neighborhood listservs.
Pre-assignment Details: Since this is a dyad study, enrollment is reported at the individual level. A total of 41 dyads (82 individuals: 41 mothers and 41 infants) consented, enrolled, and started. One dyad (2 individuals) withdrew prior to analysis, resulting in 40 dyads (80 individuals) with baseline and outcome data.
Groups:
- Diet Beverage Exposure (Mother): Mothers in the dyad were asked to ingest 20 ounces of a commercially-available diet beverage sweetened with sucralose and acesulfame-potassium.
- Diet Beverage Exposure (Infant): Infants in the dyad.
Period: Overall Study
Arm/Group | Diet Beverage Exposure (Mother) | Diet Beverage Exposure (Infant)
Started | 41 | 41
Completed | 40 | 40
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline maternal data were collected at the clinical research unit, including vital signs, height, weight, and questionnaires on medical and lactation history and lifestyle factors. Baseline infant data included length, weight, head circumference measured by research staff, and sex, gestational age, and health conditions reported by the mother.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diet Beverage Exposure (Mother) | Diet Beverage Exposure (Infant) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years, months] — Population: The columns presented separately report age for mothers (n=40) and infants (n=40), each subgroup representing half of the total participants. Therefore, the number analyzed in each column differs from the overall total to reflect the specific subgroup for which the measure applies.
  years, months
    Age | 32.4 (4.9) | 2.9 (1.6) | 17.65 (3.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The column presented separately report sex for mothers (n=40) and infants (n=40), each subgroup representing half of the total participants. Therefore, the number analyzed in each column differs from the overall total to reflect the specific subgroup for which the measure applies.
  Participants
    Sex: Female | 40 | 22 | 62
    Sex: Male | 0 | 18 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The column display race separately for mothers (n=40) and infants (n=38), with each subgroup representing participants within the dyads. The differing numbers analyzed in each column reflect the specific subgroup relevant to the measure. The lower infant count is due to two mothers choosing not to report their infant's race and/or ethnicity.
  Participants
    Race: number analyzed (Participants) | 40 | 38 | 78
    Race: White | 19 | 17 | 36
    Race: Black | 12 | 11 | 23
    Race: Asian | 2 | 0 | 2
    Race: American Indian or Alaskan Native | 1 | 1 | 2
    Race: More than one race | 6 | 9 | 15
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Baseline Sucralose Concentration in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured immediately prior to ingestion of the diet beverage containing sucralose and acesulfame-potassium.
Time Frame: Day 0 (immediately prior to diet beverage ingestion)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 0.19 (0.57)

2. Primary Outcome: 1-hour Sucralose Concentration in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 1 hour after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 1 hour post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 0.48 (0.6)

3. Primary Outcome: 2-hour Sucralose Concentrations in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 2 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 2 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 1.67 (0.98)

4. Primary Outcome: 3-hour Sucralose Concentrations in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 3 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 3 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 3.23 (1.5)

5. Primary Outcome: 4-hour Sucralose Concentrations in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 4 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 4 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 4.76 (1.99)

6. Primary Outcome: 6-hour Sucralose Concentrations in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 6 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 6 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 6.61 (2.81)

7. Primary Outcome: 8-hour Sucralose Concentrations in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 8 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 8 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 6.74 (2.76)

8. Primary Outcome: 12-hour Sucralose Concentrations in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 12 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 12 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 5.18 (2.37)

9. Primary Outcome: 24-hour Sucralose Concentrations in Breast Milk
Description: Mean concentration of sucralose in breast milk collected from mothers measured 24 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 24 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 2.24 (1.28)

10. Primary Outcome: Baseline Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured immediately prior to ingestion of the diet beverage containing sucralose and acesulfame-potassium.
Time Frame: Day 0 (immediately prior to diet beverage ingestion)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 18.11 (49.04)

11. Primary Outcome: 1-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 1 hour after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 1 hour post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 115.27 (101.52)

12. Primary Outcome: 2-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 2 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 2 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 294.22 (285.44)

13. Primary Outcome: 3-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 3 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 3 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 380.65 (327.21)

14. Primary Outcome: 4-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 4 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 4 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 405.75 (287.77)

15. Primary Outcome: 6-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 6 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 6 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 323.14 (216.90)

16. Primary Outcome: 8-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 8 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 8 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 205.91 (134.98)

17. Primary Outcome: 12-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 12 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 12 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 81.01 (59.62)

18. Primary Outcome: 24-hour Acesulfame-potassium Concentrations in Breast Milk
Description: Mean concentration of acesulfame-potassium in breast milk collected from mothers measured 24 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 24 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 28.17 (122.52)

19. Primary Outcome: Baseline Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured immediately prior to ingestion of the diet beverage containing sucralose and acesulfame-potassium.
Time Frame: Day 0 (immediately prior to diet beverage ingestion)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 0.64 (1.7)

20. Primary Outcome: 30-min Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 30 minutes after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 30 minutes post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 38.03 (15.02)

21. Primary Outcome: 1 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 1 hour after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 1 hour post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 80.25 (25.86)

22. Primary Outcome: 1.5 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 1 hour and 30 minutes after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 1.5 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 90.45 (29.14)

23. Primary Outcome: 2 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 2 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 2 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 90.59 (29.6)

24. Primary Outcome: 3 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 3 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 3 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 75.85 (28.45)

25. Primary Outcome: 4 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 4 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 4 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 57.72 (25.52)

26. Primary Outcome: 6 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 6 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 6 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 31.28 (12.82)

27. Primary Outcome: 8 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 8 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 8 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 18.31 (6.87)

28. Primary Outcome: 12 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 12 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 12 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 8.31 (1.76)

29. Primary Outcome: 24 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 24 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 24 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 5.91 (2.87)

30. Primary Outcome: 48 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 48 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 48 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 3.61 (2.30)

31. Primary Outcome: 72 Hour Sucralose Concentration in Maternal Plasma
Description: Mean concentration of sucralose in plasma collected from mothers measured 72 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 72 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 2.77 (2.28)

32. Primary Outcome: Baseline Acesulfame-potassium Concentrations in Maternal Plasma
Description: as for outcome 19
Time Frame: Day 0 (immediately prior to diet beverage ingestion)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 3.93 (11.62)

33. Primary Outcome: 30 Min Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 30 minutes after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 30 minutes post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 192.2 (80.38)

34. Primary Outcome: 1 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 1 hour after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 1 hour post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 308.98 (115.8)

35. Primary Outcome: 1.5 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 1 hour and 30 minutes after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 1.5 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 348.84 (102.77)

36. Primary Outcome: 2 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 2 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 2 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 355.69 (95.86)

37. Primary Outcome: 3 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 3 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 3 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 290.56 (72.99)

38. Primary Outcome: 4 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 4 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 4 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 203.23 (56.42)

39. Primary Outcome: 6 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 6 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 6 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 106.05 (39.44)

40. Primary Outcome: 8 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 8 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 8 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 58.09 (26.41)

41. Primary Outcome: 12 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 12 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 12 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 20.91 (6.44)

42. Primary Outcome: 24 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 24 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 24 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 5.26 (17.2)

43. Primary Outcome: 48 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 48 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 48 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 8.44 (22.82)

44. Primary Outcome: 72 Hour Acesulfame-potassium Concentrations in Maternal Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from mothers measured 72 hours after ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: 72 hours post-ingestion
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Mother)
Number analyzed (Participants) | 40
ng/ml | 8.16 (15.72)

45. Primary Outcome: Sucralose Concentrations in Infant Plasma
Description: Mean concentration of sucralose in plasma collected from infants at a single time point following maternal ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: At one of five prespecified intervals post maternal diet beverage ingestion: 1.5-3 hours, 3-5 hours, 5-7 hours, 7-9 hours, or 9-14 hours.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Infant)
Number analyzed (Participants) | 40
ng/ml | 5.0 (7.1)

46. Primary Outcome: Acesulfame-potassium Concentrations in Infant Plasma
Description: Mean concentration of acesulfame-potassium in plasma collected from infants at a single time point following maternal ingestion of a diet beverage containing sucralose and acesulfame-potassium.
Time Frame: as for outcome 45
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Diet Beverage Exposure (Infant)
Number analyzed (Participants) | 40
ng/ml | 9.2 (14.8)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collected continuously throughout the entire 10-day study period for all enrolled participants in both mother and infant groups.
Description: Adverse events were systematically monitored and assessed for all participants including both mothers and infants. No adverse events, serious or non-serious, were observed or reported during the study period.
Groups:
- Diet Beverage Exposure (Mother-Infant Dyads): Each enrolled unit is a mother-infant dyad. Mothers consume 20 oz of a commercially available diet cranberry juice sweetened with sucralose and acesulfame-potassium (ace-K).
Arm/Group | Diet Beverage Exposure (Mother-Infant Dyads)
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT05379270/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT05379270/SAP_001.pdf